CLINICAL TRIAL: NCT04160416
Title: mXELOXIRI Combined With Molecular Targeted Drug as First-line Therapy in Patients With Initially Unresectable Metastatic Colorectal Cancer: A Phase II, Single-arm, Prospective Clinical Study
Brief Title: mXELOXIRI Combined With Molecular Targeted Drug in mCRC
Acronym: TRICAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Weiqin Jiang,MD, Associate chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRICAP
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Unresectable Metastatic Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- mXELOXIRI (Experimental): Induction therapy is followed by the maintenance therapy. Induction treatment: XELOXIRI+CET/BEV Administered for 6 cycles (a maximum of 8 cycles).Bevacizumab (BEV): 5mg/kg (d.i.v.); Cetuximab 500mg/sq.m (d.i.v.)；Oxaliplatin (OX): 68 mg/sq.m (d.i.v.) Irinotecan (IRI):135 mg/sq.m (d.i.v.) CAP 1,600 mg/sq.m /day (p.o. day1-10) Administered every 2 weeks.
  Maintenance treatment: CAP+CET/BEV. The following CAP+BEV/CET therapy will be repeated in 2-week cycles.
  Interventions: Drug: Capecitabine-Oxaliplatin-Irinotecan Combination

INTERVENTIONS:
Drug: Capecitabine-Oxaliplatin-Irinotecan Combination — CAP 1,600 mg/sq.m /day (p.o. day1-10) D1-10; Oxaliplatin (OX): 68 mg/sq.m (d.i.v.) D1; Irinotecan (IRI):135 mg/sq.m (d.i.v.) D1; BEV: 5mg/kg (d.i.v.) D1; CET: 500 mg/sq.m (d.i.v.) D1; Administered every 2 weeks.

SUMMARY:
The objective is to evaluate the efficacy and safety of modified XELOXIRI combined with molecular targeted drug as first-line therapy in patients with metastatic colorectal cancer (mCRC)

DETAILED DESCRIPTION:
It is an investigator-initiated, single institution, prospective, single-arm clinical study to evaluate the efficacy and safety of modified XELOXIRI combined with molecular targeted drug as first-line therapy in patients with unresectable mCRC. Eligible patients will receive 8 cycles of mXELOXIRI with cetuximab or bevacizumab and then the maintenance therapy until disease progression (PD) or unacceptable toxicity, whichever occurs first. Study evaluation time is defined as up to 16 weeks after the first dosing of the last patient.

ELIGIBILITY:
Inclusion Criteria:

1. Personal written informed consent is obtained after the study has been fully explained
2. Histologically confirmed colon or rectal adenocarcinoma

   *Excluding appendix cancer and anal canal cancer
3. Clinically unresectable
4. Borderline resectable liver metastases of colorectal cancer considered to have poor-risk disease not deemed to be suitable for upfront resection if they had one or more of the following features assessed by a local multidisciplinary team: more than four metastases, location and distribution of metastatic disease within the liver unsuitable for resection with clear margins (e.g. involvement of both lobes of liver, invasion of intrahepatic vascular structures), extent of liver involvement precluding resection with adequate post-resection residual liver parenchyma volume for viable liver function in the immediate postoperative period, and inability to retain adequate vascular inflow and outflow to maintain viable liver function.
5. Age at enrollment is >= 20 and <= 75 years
6. Life expectancy of at least 12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1
8. Vital organ functions meet the following criteria within 14 days before enrollment.

If multiple test results are available in that period, the results closest to enrollment will be used. No blood transfusions or hematopoietic factor administration will be permitted within 2 weeks before the date on which measurements are taken.

i. Absolute neutrophil count (ANC): ≥3,000 /cu.mm ii. Platelet count: ≥10.0 × 104/cu.mm iii. Hemoglobin concentration: ≥8.0 g/dL iv. Prothrombin time (PT), activated partial thromboplastin time(APTT): ≤1.5 times upper limit of normal (ULN) v. Total bilirubin: ≤1.5 times ULN (≤3 times ULN for metastases to liver).Aspartate aminotransferase (AST), Alanine aminotransferase (ALT): ≤2.5 times ULN (≤5 times ULN for metastases to liver).

vi. Serum creatinine: ≤1.5 times ULN, or creatinine clearance: ≥30 mL/min

Exclusion Criteria:

1. Previous chemotherapy for other malignancies
2. Clinically resectable
3. Major surgical procedure within 28 days prior to study treatment initiation (such as open chest, laparoscopy, thoracoscopic surgery, laparoscopic surgery), unless only colostomy is performed; open biopsy or suturing for major trauma within 14 days of study treatment initiation; or planned major surgical procedure during the study (open chest, laparoscopy) ("major surgical procedures" does not include central venous (CV) port insertion)
4. Have received any experimental therapy (such as take part in another clinical study) within 4 weeks before treatment;
5. Receiving immunotherapy, chemotherapy, radiotherapy (except palliative radiotherapy), or hormonotherapy, which are not included in study protocol;
6. Untreated brain metastases, spinal cord compression, or primary brain tumor;
7. Pregnant, breastfeeding, positive pregnancy test (women who have menstruated in the last year will be tested), or women who are unwilling to use contraception; men who are unwilling to use contraception during the study
8. Any of the following comorbidities i. Uncontrolled hypertension ii. Uncontrolled diabetes mellitus iii. Uncontrolled diarrhea iv. Peripheral sensory neuropathy (≥Grade 1) v. Active peptic ulcer vi. Unhealed wound (except for suturing associated with implanted port placement) vii. Other clinically significant disease (such as interstitial pneumonia or renal impairment)
9. Subjects with known allergy to the study drugs or to any of its excipients.
10. Any indication of contraindications to chemotherapy;
11. Other active malignancies (synchronous malignancies, and asynchronous malignancies separated by a 5-year disease-free interval) (excluding malignancies that are expected to be completely cured, such as intramucosal carcinoma and carcinoma in situ)
12. Patients are receiving CYP3A4 strong inducer, including but not limited to aminoglutethimide, bexarotene, bosentan, carbamazepine, dexamethasone, efavirenz, fosphenytoin, griseofulvin, modafinil, nafcillin, nevirapine, oxcarbazepine, phenobarbital, diphenylhydantoin, primidone, rifabutin, rifampicin, rifapentine, hypericum perforatum;
13. The investigator judges that patients can not finish the clinical study due to medical, social, or psychological reasons, or can not sign a valid informed consent;
14. Patients with parenchymal organ transplantation who need to receive immunosuppressive therapy;
15. Evidence of HIV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 36 months
  Overall response rate
PFS | Up to 18 months
  Progression-free survival
R0 rate | Up to 18 months
  resection rate
OS | Up to 36 months
  Overall Survival
Incidence of adverse events | Up to 36 months
  Adverse events were evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. All adverse events was collected in duration from starting treatment to whichever shorter "after 30 days from withdrawal treatment" or "later treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No